CLINICAL TRIAL: NCT03294876
Title: Investigating Recovery of the Hypothalamus-pituitary-adrenal Axis in Patients With Rheumatoid Arthritis Following Exposure to Prednisolone
Brief Title: Rheumatoid Arthritis Adrenal Recovery Study
Acronym: RAAR
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC17080
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis; Adrenal Insufficiency
Keywords: Glucocorticoid; HPA axis
MeSH Terms: conditions — Arthritis, Rheumatoid; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Blood for DNA Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cortisol is a naturally occurring stress hormone, made by the adrenal glands in response to hormones produced by the pituitary and hypothalamus. Man-made forms of cortisol ('steroids', for example prednisolone) have been used for the treatment of rheumatoid arthritis since the 1950s; they are very effective at reducing inflammation.

A normal response to taking steroid treatment is that the body needs to make less cortisol. Following treatment with steroids, the system responsible for making cortisol can be slow to wake up. If someone does not make enough cortisol, they are less able to deal with stress and are at increased risk of becoming unwell, or suffering a potentially fatal adrenal crisis. It is not clear how common failure of recovery of the adrenal axis is, how long it can last for or, if any factors might predict which patients are most at risk.

This study aims to improve our understanding of hypothalamus-pituitary-adrenal (HPA) axis recovery in patients with rheumatoid arthritis treated with prednisolone. The investigators will also test potential predictive biomarkers of recovery.

The study will be conducted in hospital and a clinical research facility. Participants will undergo two visits for blood tests and will also be asked to supply three samples of saliva on six days over the three weeks of the study.

A better understanding of the physiology of HPA axis recovery should inform the development of tools which would allow prediction of patients at risk following withdrawal of steroid treatment. Such tools would be useful to improve patient safety.

DETAILED DESCRIPTION:
Cortisol is a naturally occurring stress hormone. It is made by the adrenal glands in response to hormones produced by the pituitary and hypothalamus. Man-made forms of cortisol ('steroids', for example prednisolone) have been used for the treatment of rheumatoid arthritis since the 1950s; they are very effective at reducing inflammation. Steroids are prescribed for a wide variety of inflammatory conditions. The British prevalence of chronic (greater than 3 months) steroid prescription is 1%.

A normal response to taking steroid treatment is that the body needs to make less cortisol. Following treatment with steroids, the system responsible for making cortisol (known as the hypothalamic pituitary adrenal axis (HPA axis)) can be slow to re-establish production. If someone does not make enough cortisol, they are less able to deal with stress and are at increased risk of becoming unwell, or suffering a potentially fatal adrenal crisis. The prevalence of inadequate cortisol production following treatment with steroids is between 10-30% of patients; its duration and whether any patient factors might predict which patients are at risk is unclear. Generally studies have been small in size and do not report sufficient information to determine if any potential factors maybe useful predictors; for example age, sex, length of treatment, length of time off treatment, other medications.

Rheumatoid arthritis (RA) has a prevalence of 1%. Patients are usually treated with a 13 week course of prednisolone in a reducing dose (treatment regimen known as COBRA-light) at diagnosis. 1-2 patients present each week to the rheumatology department in Edinburgh with a new diagnosis of RA. At the end of the initial COBRA-light treatment, the adrenal axis is not routinely assessed in these patients. It is assumed that the slow reducing dosage of steroids reduces the risk of ongoing adrenal insufficiency. It should be noted that the meta-analysis of Joseph et al. demonstrated weaning had little impact upon the recovery of the HPA axis. These patients are thus potentially at risk of the morbidity and mortality associated with an underactive HPA axis.

This study aims to improve our understanding of HPA axis recovery in patients with rheumatoid arthritis following treatment with prednisolone. The investigators will also test two novel potential predictive biomarkers of recovery.

A better understanding of the physiology of HPA axis recovery should inform the development of tools which would allow prediction of patients at risk following withdrawal of steroid treatment. Such tools would be useful to improve patient safety and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis
* Treatment with prednisone via COBRA light regime
* Age over 18

Exclusion Criteria:

* Adrenal or pituitary disease
* Alcohol intake over 21 units/week
* Shift work (night shifts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited following 13 week weaning dose of prednisone for treatment of early arthritis
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Synacthen test 1 | Day 1
  Short synacthen test the after withdrawal of prednisone
Synacthen test 2 | Day 21
  Short synacthen test 21 days after withdrawal of prednisone
Cortisol awakening curve | 2 days in each of weeks 1, 2 and 3
  Salivary cortisol at waking, and 30 mins and 45 mins after waking

SECONDARY OUTCOMES:
Single Nucleotide Polymorphism | Assessed at day 0
  Assessment of an SNP as a predictor of prolonged HPA axis suppression
Quality of life | Assessed at day 21
  SF-36 (Short Form Survey) assessed quality of life
Metabolite panel | Day 0
  Assessment of a panel of metabolites which might predict HPA suppression

CONTACTS AND LOCATIONS:
Overall Officials: Thomas JG Chambers, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Metabolic Unit, Western General Hospital, NHS Lothian, Crewe Road, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No